CLINICAL TRIAL: NCT04412135
Title: The Point of View of Hematological Cancer Patients and Their Loved Ones Regarding Spirituality During the Initial Healing Phase
Brief Title: The Point of View of Hematological Cancer Patients and Their Loved Ones Regarding Spirituality
Acronym: SPIRIHEMATO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0050
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-03

CONDITIONS: Hematologic Cancer
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Spiritual Therapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: spirituality — Patients will take three questionnaires (FACIT-Sp, Euroqol 5 dimensions and ESAS)

SUMMARY:
The management of patients with malignant hemopathy is based on comprehensive management. In this context and faced with the various difficulties encountered by cancer patients, the question of spirituality and its experience is central. Spirituality refers to the person's attachment to what inspires and gives him foundation, as well as the beliefs, values, and existential experiences associated with it, whether these are religious in nature or not. Although the concept has been identified as a resource in the literature and widely treated in an end-of-life context, assessing the needs of patients with hematological cancer and their loved ones in terms of spirituality from the initiation of treatment does not has not been developed

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years with a recent diagnosis of hematological cancer (lymphoma or leukemia) and in treatment;
* Patients who speak and read French;
* Patients in general condition (physical and mental) judged emotionally and physically fit by the referring nurse to answer the questionnaires;
* Patients benefiting from a social security scheme,
* Patients who signed the non-objection form after being informed of the study,

family person:

* Have been designated by the patient as being the loved one they wish to include with them;
* Aged ≥ 18 years;
* Fluent in and reading French;
* Having signed the non-objection form after being informed of the study.

Exclusion Criteria:

* Patients in recurrence / progress or in remission of cancer;
* Patients in the terminal phase of the disease.

Family person:

person in the curative phase of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hematologic cancer patient and family member
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
FACIT-Sp questionnaire | 15 minutes

IPD SHARING:
Plan to Share IPD: No